CLINICAL TRIAL: NCT04643574
Title: Pilot Study to Assess the Feasibility, Safety and Efficacy of Adoptive Transfer of Autologous Tumor-Infiltrating Lymphocytes Enriched for Tumor Antigen Specificity (NeoTIL) in Advanced Solid Tumors
Brief Title: NeoTIL in Advanced Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Principal Investigator, Dr Blanca Navarro-Rodrigo, MD, MD, Centre Hospitalier Universitaire Vaudois
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHUV-D0-0018-NeoTIL-2019
Record Dates: First submitted 2020-11-17; First posted 2020-11-25 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Solid Tumor, Adult
MeSH Terms: interventions — neotil; Cyclophosphamide; fludarabine; Interleukin-2; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- NeoTIL-ACT + LDI (Experimental): Non-myeloablative lymphodepleting chemotherapy (fludarabine and cyclophosphamide), Low Dose Irradiation (LDI), ex vivo expanded Tumor Infiltrating Lymphocyte (TIL), enriched for tumor antigen specificity (NeoTIL)-Adoptive Cell Therapy (ACT), Interleukin-2 (IL-2).
  Interventions: Biological: NeoTIL; Drug: Cyclophosphamide; Drug: Fludarabine; Drug: Interleukin-2; Radiation: Radiotherapy

INTERVENTIONS:
Biological: NeoTIL — Adoptive transfer of ex vivo expanded Autologous Tumor-Infiltrating Lymphocytes enriched for tumor antigen specificity (NeoTIL)
Drug: Cyclophosphamide — Cyclophosphamide will be administered as an intravenous (IV) infusion for two days.
Drug: Fludarabine — Fludarabine will be administered as an intravenous (IV) infusion for five days.
Drug: Interleukin-2 — After TIL infusion, IL-2 (optional) will be started as a bolus administration every eight hours, for a maximum of fourteen doses.
Radiation: Radiotherapy — Low-dose irradiation (1Gy) will be administered using tomotherapy to tumor lesions once before NeoTIL infusion.

SUMMARY:
Single center, single arm pilot trial to test the feasibility, safety and efficacy of NeoTIL-ACT combined with low-dose irradiation (LDI) in patients with advanced, recurrent or metastatic solid tumors.

The trial is based on lymphodepleting chemotherapy followed by LDI, and then ACT utilizing ex vivo expanded TIL, enriched for tumor antigen specificity (NeoTIL), in combination with high dose Interleukin-2 (IL-2) (optional, depending on patient's tolerance).

LDI will be administered once to metastatic lesions using tomotherapy.

DETAILED DESCRIPTION:
The objective of the trial is to define the feasibility, safety, and efficacy of NeoTIL-ACT in combination with LDI in patients with advanced, recurrent or metastatic solid tumors, as categorized in two molecularly defined cohorts.

Study treatment will begin with intravenous (IV) non-myeloablative (NMA) lymphodepleting chemotherapy composed by fludarabine and cyclophosphamide. Both treatments will be started on the same day. Fludarabine will be administered from for five days, and cyclophosphamide ffor two days. Low-dose irradiation (LDI) will be administered once, to tumor lesions using tomotherapy.

Patients will receive NeoTIL infusion intravenously followed by high dose IL-2 administration every eight hours, for a maximum of fourteen doses. Supportive care will be given as needed during the whole treatment period.

Patients achieving a stable disease, partial response or complete response after NeoTIL-ACT treatment will then enter a clinical follow-up period for 5 years.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with advanced (not radically treatable), recurrent or metastatic solid tumors of any histology with the exception of primary central nervous system tumors, who have received, and then progressed or been intolerant to at least one standard therapy regimen in the advanced or metastatic setting if such a therapy exists, and have been considered for all other potentially efficacious therapies prior to enrollment. If the participant refuses, or is not eligible for these regimens in the opinion of the investigator, the reason must be documented in the medical record.
2. Patients who have previously undergone tumor resection or biopsy and for whom pre-Rapid Expansion Protocol (REP) NeoTIL cultures are ongoing or completed.
3. At least one lesion accessible to biopsy for translational research (TR) at baseline and D30, without putting the patient at unusual risk.
4. Male or female age ≥ 18 to ≤ 70 years at the time of informed consent. Patients aged >70 will be evaluated by the investigator, and decision will be made according to patient's status, upon agreement with the PI.
5. Clinical performance status of Eastern Cooperative Oncology Group (ECOG) of 0 to 2.
6. Life expectancy of greater than 12 weeks.
7. Radiologically measurable disease (as per Response Evaluation Criteria in Solid Tumours [RECIST] v1.1).

   1. Modified RECIST should be used for mesothelioma
   2. Prostate Cancer Working Group 3 (PCWG3) criteria should be used for prostate cancer
8. Adequate serology defined by the following laboratory results:

   1. Negative test for Human Immunodeficiency Virus (HIV)
   2. Patients with active or chronic hepatitis B (defined as having a positive hepatitis B surface antigen [HBsAg] test at pre-screening) are not eligible.

      * Patients with past/resolved Hepatitis B virus (HBV) infection (defined as having a negative HBsAg test and a positive antibody to hepatitis B core antigen (anti-HBc) antibody test) are eligible, if HBV deoxyribonucleic acid (DNA) test is negative.
      * HBV DNA must be obtained in patients with positive hepatitis B core antibody prior start of study treatment.
   3. Patients with active hepatitis C are not eligible. Patients positive for Hepatitis C virus (HCV) antibody are eligible only if polymerase chain reaction (PCR) is negative for HCV ribonucleic acid (RNA).
9. Hematology

   1. Absolute neutrophil count ≥ 1.0 x 109 cell/L without the support of granulocyte colony stimulating factor (G-CSF).
   2. Platelet count ≥ 100 x109 cell/L
   3. Hemoglobin ≥ 80 g/L. Subjects may be transfused to reach this cut-off.
10. Coagulation

    a. International normalization ratio (INR) ≤1.5 times the upper limit of normal (x ULN) unless the subject is receiving anticoagulant.

    i) Exception: for patients with hepatocellular carcinoma (HCC), the INR may be up to 2.2, as long as the Child-Pugh score is A6 maximum.

    b. Partial thromboplastin time (PTT) or activated partial thromboplastin time (aPTT) ≤ 1.5 x ULN unless the subject is receiving anticoagulant therapy.
11. Chemistry:

    1. Serum alanine transaminase (ALT) / aspartate aminotransferase (AST) ≤ to 3 x ULN i) Exception: ALT/AST considered related to liver metastasis ≤ to 5 x ULN ii) Exception: for patients with HCC serum ALT/AST ≤ to 5 x ULN
    2. Total bilirubin ≤1.5 x ULN i) Exception: in patients with Gilbert's syndrome who must have a total bilirubin ≤2.5 x ULN ii) Exception: total bilirubin considered related to liver metastasis ≤3 x ULN iii) Exception: for patients with HCC total bilirubin ≤2.3 x ULN, as long as the Child-Pugh score is A6 maximum
    3. Creatinine clearance by Cockcroft-Gault formula ≥ 40 ml/min
12. Adequate cardiovascular function, with documented left ventricular ejection fraction (LVEF) ≥ 45%. This parameter must be documented within 12 weeks before registration
13. Adequate respiratory function with forced expiratory volume in 1 second (FEV1) ≥ 50% predicted, forced vital capacity (FVC) ≥ than 50% predicted and diffusing capacity for carbon monoxide (DLCO) ≥ than 50% predicted corrected. Patients with lung cancer or mesothelioma and values slightly under these limits (but >30% of predicted) can be enrolled after discussion and approval by the PI. These parameters must be documented within 12 weeks before registration
14. At the time the patient receives the NMA chemotherapy regimen (D-7):

    1. ≥14 days or 5 half-lives must have elapsed from any chemotherapeutic cytotoxic drug, whichever is shorter.
    2. ≥28 days must have elapsed from bevacizumab, aflibercept and other anti-angiogenic antibodies
    3. ≥28 days or 5 half-lives (whichever is shorter) must have elapsed from a non-cytotoxic drug including but not limited to trastuzumab, pertuzumab, and other molecular targeted therapy (such as tyrosine kinase inhibitors, etc…) i) Note: In case of probable tumor flare upon stopping of the non-cytotoxic drug, the investigator may decide to shorten this delay, upon agreement of the Principal Investigator (PI), in a case-by-case approach.
    4. ≥21 days must have elapsed from the last antibody therapy that could affect an anti-cancer immune response, including but not limited to anti-Cytotoxic T-lymphocyte-associated protein 4 (CTLA4), anti-Programmed cell death protein 1 (PD-1), anti-Programmed death-ligand 1 (PD-L1), anti-Tumor Necrosis Factor Receptor Superfamily, member 4 (OX-40), or anti-Lymphocyte-activation gene 3 (LAG3) antibody therapy or their combination
    5. Exceptions: denosumab and biphosphonates are permitted (and will be administered as standard of care [SOC]).
    6. Exceptions: androgen-deprivation therapy (ADT) for prostate cancer and hormonal therapy for breast cancer are permitted (and will be administered as SOC).
15. Patients' toxicities from previous therapies must have recovered to at least grade 1 according to National Cancer Institute Common Terminology Criteria for Adverse v5.0 (NCI CTCAE v5.0), except for toxicities described below, as long as they do not put at risk the patient's condition and do not require systemic immunosuppressive steroids at immunosuppressive doses, including but not limited to:

    * Fatigue
    * Alopecia
    * Skin disorders
    * Stable neuropathy
    * Endocrinopathies requiring replacement treatment Note: For other medical conditions, or for any other toxicity with a higher grade but controlled by adequate treatment, prior discussion and agreement with the PI is mandatory.

    Note: Patients may have undergone surgical procedures within the past 3 weeks, as long as all toxicities have recovered to grade 1 or less.
16. For women of childbearing potential (WOCBP: sexually mature women who have not undergone a hysterectomy and/or bilateral oophorectomy, have not been naturally post-menopausal for at least 12 consecutive months or have a serum follicle-stimulating hormone (FSH) < 40 milli-International Unit [mIU]/ml):

    1. Agreement to follow instructions for method(s) of contraception for the couple, from screening until month 6 post start of NMA chemotherapy of the study.
    2. Negative pregnancy test (urine or serum) during screening
17. For men participating in the trial and their female partners: agreement to follow instructions for method(s) of contraception for the couple from screening until month 6 post start of NMA chemotherapy of the study.

Exclusion Criteria:

1. Patients with an active second malignancy, except for

   1. non-melanoma skin cancer that has been apparently cured or successfully resected
   2. carcinoma in situ as long as they have been adequately treated
   3. Any malignancy that can be adequately managed expectantly without compromising prognosis, and after PI agreement.

   Patients who have a history of malignancy are not considered to have an active malignancy if they have completed therapy since at least 2 years and are considered by their treating investigator to be at ≤ 30% risk for relapse.
2. Patients with symptomatic and/or untreated brain metastases. Patients with definitively-treated brain metastases will be considered for enrollment after agreement with PI, as long as lesions are stable for ≥ 14 days prior to beginning the chemotherapy, there are no new brain lesions, and the patient does not require ongoing corticosteroid treatment.
3. Patients with known peritoneal metastases who have a recent history of intermittent bowel obstruction (even partial), unless such obstruction has been resolved. Agreement with the PI is mandatory.
4. Patients with leptomeningeal carcinomatosis
5. History of idiopathic pulmonary fibrosis or evidence of active pneumonitis (any origin)
6. History of recent myocardial infarction or unstable angina, either within six months of enrolment
7. Documented Child-Pugh score of B or C for hepatocellular carcinoma patients with known underlying liver dysfunction
8. Active severe systemic infections within four weeks prior to beginning of NMA chemotherapy.
9. Patient requiring regular systemic immunosuppressive therapy (for example for organ transplantation, chronic rheumatologic disease); all immunosuppressive medications including but not limited to steroids, mycophenolate mofetil, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor-alpha (TNF-alpha) agents must have been discontinued within the last two weeks prior to starting NMA chemotherapy.

   1. Note: Use of inhaled or topical steroids or corticosteroid use for radiographic procedures is permitted
   2. Note: The use of physiologic corticosteroid replacement therapy is permitted.
10. History of severe immediate hypersensitivity reaction to any of the agents used in this study.
11. Women who are pregnant or breastfeeding because of the potentially dangerous effects of the treatment on the fetus or infant.
12. Subjects for whom there are concerns that they will not reliably comply with the requirements for contraception should not be enrolled into the study.
13. Any serious underlying medical condition that could interfere with study medication and potential adverse events.
14. Any mental or other impairment that may compromise compliance with the requirements of the study.
15. Patient participation in any other study currently receiving treatment. If the patient is in the follow-up period, he/she may be enrolled, as far as the elapsed time since the last previous treatment administration and the preparative regimen (NMA chemotherapy) is respected according to Inclusion Criteria n°14.
16. Participation in a research project using radiation sources exceeding an effective dose of 5 millisievert (mSv) with no direct benefit within the 12 last months.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2021-03-09 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the number of patients who successfully receive NeoTIL-ACT in combination with LDI (feasibility) | Evaluated for each patient at day 0
  Defined as:
  * Planned NMA chemotherapy regimen
  * Planned LDI
  * At least partial NeoTIL infusion
  * No minimum IL-2 requirement
Toxicity of NeoTIL-ACT in combination with LDI | Treatment limiting toxicity (TLT) period: from day starting NMA chemotherapy to day 30 post NeoTIL infusion
  Number of patients with adverse events as assessed by CTCAE version 5.0
Objective response rate (ORR; efficacy of NeoTIL-ACT in combination with LDI) | Up to 6 months
  Defined as best overall response (complete response or partial response) across all assessment time points, according to RECIST 1.1, mRECIST for mesothelioma or PCWG3 for prostate cancer

SECONDARY OUTCOMES:
Disease Control Rate (DCR) | 1, 3, 6, 9,12 months
  Achievement of complete response, partial response or stable disease
Objective response rate (ORR) | 1, 3, 6, 9, 12 months
  Best overall response
Progression free survival (PFS) | 5 years
  Time from enrollment until objective tumor progression or death
Overall survival (OS) | 5 years
  Time from enrollment until death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Blanca Navarro-Rodrigo, MD, PhD, Principal Investigator — Centre Hospitalier Universitaire Vaudois; George Coukos, MD, PhD, Study Chair — Centre Hospitalier Universitaire Vaudois
Locations (1):
- centre hospitalier universitaire vaudois (CHUV), Lausanne, Canton of Vaud, Switzerland